CLINICAL TRIAL: NCT02100644
Title: Valproate Dose Reduction and Its Clinical Evaluation by Introducing Lamotrigine in Japanese Women With Epilepsy - Single Arm, Multicenter, and Open-label Study -
Brief Title: Valproate Dose Reduction and Its Clinical Evaluation by Introducing Lamotrigine in Japanese Women With Epilepsy - Single Arm, Multicenter, and Open-label Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200776
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamotrigine (Experimental): The study objective is to examine whether the VPA dose can be reduced by additional administration of LTG in Japanese pre-menopausal female epilepsy patients, whose seizures are well controlled by VPA monotherapy. Then VPA is the standard product in this stuudy, not the investigational product.
  Interventions: Drug: Lamotrigine tablets 25/100 mg

INTERVENTIONS:
Drug: Lamotrigine tablets 25/100 mg — Lamotrigine (LTG) is administered according to the package insert: that is, 25 mg of LTG will be orally administered once every other day for the first 2 weeks and then once daily for the next 2 weeks. Thereafter, the dose will be gradually escalated by 25-50 mg every 1-2 week for once or twice daily administration. During the VPA reduction phase and LTG&VPA maintenance phase, as specified in the information of package insert, maintenance dose of LTG will be administered twice daily.

SUMMARY:
The purpose of this study is to examine whether the VPA (Valproate) dose can be reduced by additional administration of LTG (Lamotrigine) in Japanese pre-menopausal female epilepsy patients aged 15 years or older, whose seizures are well controlled by VPA monotherapy.

DETAILED DESCRIPTION:
RATIONALE In several studies that investigated the effects of in utero exposure to AEDs (antiepileptic drugs) on fetal malformations and intellectual development in children after birth, it has been reported that VPA causes neonatal malformations and decreases intelligence of children in a dose dependent manner, whereas such a risk is low in LTG (Hernandez-Díaz et al., 2012; Meador et al., 2013). It has also been reported that LTG as adjunctive therapy with VPA is effective in inhibiting seizures in patients with poorly controlled seizures, and adverse events under VPA monotherapy can be relieved by subsequently reducing VPA dose after LTG is combined (Sale et al., 2005; Jozwiak et al., 2000; Morris et al, 2004; Buchanan, 1996). Thus, by considering the benefits of replacing VPA by LTG in childbearing women, we will examine whether VPA dose can be reduced by introducing LTG in Japanese female epilepsy patients under VPA monotherapy (aged ≥ 15 years, pre-menopausal).

STUDY DESIGN Single arm, multicenter, and open-label study TIME FRAME

* Screening(Retrospective review of medical records for 12 weeks)
* LTG escalation phase (8-18 weeks)
* VPA reduction phase (3-16 weeks)
* LTG & VPA maintenance phase (12 weeks)
* Follow up (1-4 weeks) PRIMARY OBJECTIVE To examine whether the VPA dose can be reduced by additional administration of LTG (up to 200 mg/d if there are no safety concerns) in Japanese pre-menopausal female epilepsy patients aged 15 years or older, whose seizures are well controlled by VPA monotherapy (fixed maintenance dose of 400-1200 mg/d).

SECONDARY OBJECTIVES

* To investigate the steady state concentration of LTG immediately before VPA dose reduction, at the time of VPA dose reduction, and during the LTG&VPA maintenance phase.
* To investigate the safety and tolerability associated with additional administration of LTG followed by dose reduction of VPA.

ELIGIBILITY:
Inclusion Criteria:

1. (Target disease) Epilepsy patients having the following seizure types as classified by the International Classification of Epileptic Seizures

   * Partial seizures (with or without secondary generalization)
   * Tonic-clonic seizures with or without myoclonus but without other generalized seizure type(s)
2. Subjects having a confident diagnosis of epilepsy that is uncomplicated by pseudoseizures such as psychogenic nonepileptic seizures
3. Subjects whose seizures have been controlled for 12 weeks prior to start of the investigational product with a stable maintenance dose of VPA monotherapy (400-1200 mg/d)
4. (Age and gender)

Japanese pre-menopausal women who are at least 15 years old at the time of consent, not lactating, and can agree to use any of the following types of contraception in a reliable fashion:

1. Complete abstinence during the study as well as for a period after the study to account for elimination of the investigational product (a minimum of 2 weeks)
2. Consistent and correct use of any of the following contraceptive methods

   * Surgical sterilization of male partner (i.e., male partner is the sole sexual partner for the female subject and is sterilized prior to the subject's entry into the study)
   * Intrauterine device with a failure rate of less than 1% per year
   * Double barrier method (e.g., spermicide plus a condom or a diaphragm) Note: Women who have had a hysterectomy or tubal ligation are considered to be of non-childbearing potential. Since a pharmacokinetic interaction has been observed between LTG and estrogen-based oral contraceptives, the use of hormonal therapy such as for contraception or hormone replacement therapy is not allowed.

     5.Outpatients 6.Subjects who can keep a seizure diary 7.Subjects who can understand and sign the informed consent. If the subject is under 20 years old at the time of consent, both the subject and subject's legally acceptable representative have to sign the consent to participate in the study.

     8.QTc <480 msec for subjects with bundle branch block or QTc <450 msec for other subjects, in which QTc is measured by either single or triplicate-averaged ECG 9.Subjects who can comply with dosing of the investigational and standard products and all study procedures

Exclusion Criteria:

1. Subjects with a history of hypersensitivity to LTG
2. Subjects with a history of rash associated with other AED treatments.
3. Subjects who have received another AED besides VPA during the 12 weeks prior to start of the investigational product
4. Subjects with status epilepticus during the 6 months prior to start of the investigational product
5. Subjects with a history of substance (including alcohol and drug) dependence or substance abuse as defined by the DSM-IV-TR within 12 months or 1 month, respectively, prior to start of the investigational product
6. Subjects with a severe acute or chronic illness likely to impair drug absorption, distribution, metabolism, or excretion; or subjects with any unstable physical symptom likely to require hospitalization during the study
7. Subjects with a severe psychiatric disorder that affects the procedures of the study or drug assessment
8. Subjects with an acute or progressive neurological disorder or an organic disease
9. Subjects with any clinically significant cardiac, renal, or hepatic medical condition. Any patient with these conditions will be excluded from the study even if these conditions are being controlled with a chronic therapy.
10. Subjects with an unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) Note: Chronic stable hepatitis B and C are acceptable if the subjects otherwise meet the inclusion criteria. However, the subjects with chronic stable hepatitis B will be excluded if significant immunosuppressive agents are being administered due to a risk of hepatitis B reactivation.
11. Subjects who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study
12. Subjects who are suspected to have an urea cycle disorder as below:

    * Subjects with a history of encephalopathy or coma of unknown cause
    * Subjects with a family history of infant death of unknown cause or urea cycle disorder
13. Subjects taking inducers of LTG glucuronidation (i.e., rifampicinor lopinavir/ritonavir), atazanavir/ritonavir, risperidone, or oral contraceptives or hormone drugs containing estrogen
14. Subjects taking carbapenem antibiotic (i.e., panipenem/betamipron, meropenem hydrate, imipenem hydrate/cilastatin sodium, biapenem, doripenem hydrate, or tebipenem pivoxil)
15. Subjects who have participated in other clinical studies within 3 months prior to start of the investigational product
16. Subjects who have had active suicidal plans/intent or suicidal thoughts in the past 3 months prior to start of the investigational product; or subjects who have history of suicide attempts in the last 1 year prior to start of the investigational product or of multiple suicide attempts in their lifetime
17. Subjects whom the investigator or subinvestigator considers ineligible for the study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04-12 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2015-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Japan (7):
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 200776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) receiving monotherapy treatment with sodium valproate (VPA) maintenance dose of 400-1200 milligrams/day [mg/d]) due to a history of partial seizures (including secondary generalized seizures) or tonic-clonic seizures, and whose seizures had been controlled for 12 weeks (wk) prior to start of treatment were enrolled in the study.
Pre-assignment Details: A total of 33 participants were enrolled into the study and 20 participants completed the study.
Groups:
- Escalation Phase: LTG Plus VPA: Participants received a fixed maintenance dose of VPA (400-1200 mg/d) along with lamotrigine (LTG) which was gradually escalated to 200 mg/d in accordance with the information of package insert: i.e. 25 mg of LTG was orally administered once every other day for the first 2 weeks and then once daily for the following 2 weeks. Thereafter, LTG was gradually escalated by 25 to 50 mg every 1 to 2 weeks for once or twice daily administration. If there were safety concerns, the LTG dose was decreased to 100 mg/d at the discretion of the investigator or sub-investigator. If there were still safety concerns despite the dose reduction to 100 mg/d, LTG was discontinued. The total duration of this phase was 8 to18 weeks.
- Reduction Phase: LTG Plus VPA: Participants received a range of VPA dose reduction as follows: When VPA was reduced to 300 mg/d, the range of reduction was determined at the discretion of the investigator or sub-investigator: e.g., 1000 mg/d (2 weeks), 800 mg/d (2 weeks), 600 mg/d (2 weeks), 400 mg/d (2 weeks), 300 mg/d OR 1000 mg/d (4 weeks), 600 mg/d (4 weeks), 300 mg/d and when VPA was reduced to less than 300 mg/d, the dose was reduced to 300, 200, 100, and 0 mg/d in 100 mg decrements in steps of at least one week duration. When VPA was concomitantly used, LTG was administered twice daily with 200 mg/d as a maintenance dose. If there were safety concerns during the LTG Escalation Phase, a fixed maintenance dose of 100 to 200 mg/d of LTG was administered twice daily. When VPA was withdrawn (that is, VPA was reduced to 0 mg/d), LTG was required to be increased by 50-100 mg/d. If there were any safety concern, 25 mg increment was also available. The total duration of this phase was 4 to16 weeks.
- Maintenance Phase: LTG Plus VPA: Participants received two different treatments. In one group, participants received a fixed maintenance dose of LTG 200 mg/d (or 100 to 200 mg/d if there were safety concerns during the LTG Escalation Phase) and VPA 100 mg/d (or higher if seizures occurred during the VPA Reduction Phase) were administered twice and 1-3 times daily, respectively, for 12 weeks. The frequency of administration was not changed. If seizures occurred, VPA dose could be increased/re-introduced. On the other group, after VPA was withdrawn, LTG dose was escalated up to 300 mg/d with 50-100 mg increment per 1-2 weeks. If there was safety concern or if remaining dose to 300 mg/d was below 50 mg, 25 mg increment was also available. If seizures occurred, LTG dose was increased up to 400 mg/d. If there was safety concern, LTG dose was decreased to 100 mg/d. If there was still safety concern at 100 mg/d, the participants were discontinued from the study. The total duration of this phase was 12 weeks.
Period: LTG Escalation Phase
Arm/Group | Escalation Phase: LTG Plus VPA | Reduction Phase: LTG Plus VPA | Maintenance Phase: LTG Plus VPA
Started | 33 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 13 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: VPA Reduction Phase
Arm/Group | Escalation Phase: LTG Plus VPA | Reduction Phase: LTG Plus VPA | Maintenance Phase: LTG Plus VPA
Started | 0 | 20 | 0
Completed | 0 | 20 | 0
Not Completed | 0 | 0 | 0
Period: LTG and VPA Maintenance Phase
Arm/Group | Escalation Phase: LTG Plus VPA | Reduction Phase: LTG Plus VPA | Maintenance Phase: LTG Plus VPA
Started | 0 | 0 | 20
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LTG Plus VPA (Phase 1, 2 and 3): Par. received a fixed maintenance (maint) dose of VPA (400-1200 mg/d) along with LTG gradually escalated to 200 mg/d in accordance with the package insert information: i.e. 25 mg of LTG was orally administered once every other day for the first 2 wk and then once daily for the following 2 wk. Thereafter, LTG was gradually escalated by 25 to 50 mg every 1 to 2 wk for once or twice daily administration. Par. received a range of VPA dose reduction as follows: When VPA was reduced to 300 mg/d, the range of reduction was as follows: 1000 mg/d (2 wk), 800 mg/d (2 wk), 600 mg/d (2 wk), 400 mg/d (2 wk), 300 mg/d OR 1000 mg/d (4 wk), 600 mg/d (4 wk), 300 mg/d and when VPA was reduced to < 300 mg/d, the dose was reduced to 300, 200, 100 and 0 mg/d in 100 mg decrements in steps of at least one wk duration. Par. received a fixed maint dose of LTG 200 mg/d and VPA 100 mg/d or a maint dose of LTG 200-400 mg/d were administered twice and 1-3 times daily for LTG and VPA, respectively, for 12 wk
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.6 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian- Japanese Heritage | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Reduction in Daily VPA Dose
Description: The VPA dose reduction from Baseline is defined as post VPA dose minus the Baseline VPA dose < 0. Baseline VPA dose is the dose at the Baseline visit (Week 0) and the post VPA dose is the last VPA dose during the LTG and VPA Maintenance Phase. Percentage of participants with dose reduction during the LTG and VPA Maintenance Phase is presented.
Time Frame: Baseline and at the end of the LTG and VPA Maintenance Phase, 24-46 weeks that can be varied by durations of the LTG Escalation Phase and VPA Reduction Phase
Population: Full analysis set (FAS): comprised of all participants in the Safety Population who provided at least one efficacy data after the first dose of the investigational product during the LTG Escalation Phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Percentage of participants | 60.6 [42.14 to 77.09]

2. Primary Outcome: Percent Change in the VPA Dose
Description: Percent change in VPA dose is calculated as (pre-dose - post-dose) / pre-dose x 100. Pre-dose is the VPA dose at the Baseline visit and post-dose is the last VPA dose during the LTG and VPA Maintenance Phase.
Time Frame: as for outcome 1
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Percentage of reduction
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Percentage of reduction | -60.10 (49.290)

3. Secondary Outcome: Number of Days in Total That Epileptic Seizures Occurred up to the LTG and VPA Maintenance Phase
Description: The participants with no seizure, had no record in seizure dairy. Only those participants with more than one seizure were assessed for this Outcome Measure.
Time Frame: Baseline and up to 46 weeks
Population: FAS Population
Measure: Number; unit: Days
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Days | 2

4. Secondary Outcome: Change From Baseline in Quality of Life in Epilepsy-31-P (QOLIE-31-P) in Participants Aged 18 Years and Older
Description: QOLIE-31-P is a questionnaire analyzed according to the scoring manual at Baseline, at the end of LTG/VPA Maintenance Phase and withdrawals for the participants aged 18 years and older (n=26, excluding 1 participant withdrawn due to protocol violation). Overall score was calculated as an average of sub scores that were normalized to 0 to 100. QOLIE-31-P has 7 subscale items (energy, mood, daily activities, cognition, medication effect, seizure worry and overall QOL). Higher score presents higher quality of life. Epileptic symptoms generally affect the QOL of participants, and so QOLIE-31-P is world widely used for the QOL assessment of adult participants. Baseline is defined as Day 1 (pre-dose) value. Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline and up to 46 weeks
Population: FAS Population. Only those participants available at the indicated phase were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Scores on a scale
  LTG Escalation-Withdrawal, n=10 | -7.19 (7.531)
  LTG and VPA Maintenance-Visit 5, n=16 | 0.19 (9.082)

5. Secondary Outcome: Change From Baseline in Quality of Life in Epilepsy for Adolescents (QOLIE-AD-48) in Participants Aged 15-17 Years
Description: QOLIE-AD-48 is a questionnaire analyzed according to the scoring manual at Baseline, at the end of the LTG/VPA Maintenance Phase and withdrawals for participants aged 15-17 years (n=6). Particpants who has started by QOLIE-AD-48 were using the same questionnaire even after 18 years old. Overall score was calculated as an average of sub scores that were normalized to 0 to 100. QOLIE-AD-48 has 8 subscale items (epilepsy impact, memory/concentration, physical fuctioning, stigma, social support, school behavior, attitudes towards epilepsy and health perceptions). Higher score presents higher quality of life. Epileptic symptoms generally affect the QOL of participants, and so QOLIE-AD-48 is world widely used for the QOL assessment of non-adult participants. Baseline is defined as Day 1 (pre-dose) value. Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline and up to 46 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Units on a scale
  LTG Escalation-Withdrawal, n=2 | -10.83 (11.862)
  LTG and VPA Maintenance-Visit 5, n=4 | -2.67 (6.356)

6. Secondary Outcome: Percentage of Participants Who Completed or Discontinued From the Study
Description: Following cases were considered for participants to have completed a part of or whole of the study. For whole period completion: participants who completed the last LTG and VPA Maintenance Phase visit (M5) in the LTG and VPA Maintenance Phase and follow-up examination. For LTG Escalation Phase completion: participants who reached 200 mg/d of LTG (or 100-200 mg/d of LTG if there were safety concerns) within 8-18 weeks of the phase. For VPA Reduction Phase completion: participants who completed the last fixed dose of VPA Reduction Phase visit (0 mg/d) (FR4) of the phase. For LTG and VPA Maintenance Phase completion: participants who completed M5 of the phase. Participants who met any of the withdrawal criteria after the start of investigational product were considered to have discontinued the study. Percentage of participants who completed or discontinued/withdrawn from the study is presented.
Time Frame: Up to 50 weeks
Population: Enrolled Population: comprised of all participants who had a Baseline (Week 0) visit.
Measure: Number; unit: Percentage of participants
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Percentage of participants
  Completed | 61
  Withdrawn | 39

7. Secondary Outcome: Number of Participants With Adverse Events (AEs), AEs Leading to Discontinuation of the Investigational Product and/or Withdrawal From the Study, Drug-related AEs, Deaths and Serious Adverse Events (SAEs) Throughout the Study
Description: An AE is defined as untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity, is a congenital anomaly/birth defect, based on medical or scientific judgement and all events of possible drug-induced liver injury.
Time Frame: From the start of study treatment until follow-up (up to 50 weeks)
Population: Safety Population: comprised of participants who received at least one dose of the investigational product during the LTG Escalation Phase.
Measure: Number; unit: Participants
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Number analyzed (Participants) | 33
Participants
  Any AEs | 30
  Drug-related AEs | 17
  Any SAEs | 4
  AEs leading to discontinuation/withdrawal | 9
  AEs leading to death | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment and until the follow-up contact (up to 50 weeks).
Description: AEs and SAEs were collected from participants of the safety population, comprised of all participants who received atleast one dose of the investigational product during the LTG Escalation Phase.
Arm/Group | LTG Plus VPA (Phase 1, 2 and 3)
Serious Adverse Events (participants affected / at risk) | 4/33
Other Adverse Events (participants affected / at risk) | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTG Plus VPA (Phase 1, 2 and 3) (N=33)
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTG Plus VPA (Phase 1, 2 and 3) (N=33)
Nasopharyngitis (Infections and infestations) | 9
Gastroenteritis (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Somnolence (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Seasonal allergy (Immune system disorders) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Insomnia (Psychiatric disorders) | 2
Pyrexia (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.